CLINICAL TRIAL: NCT05265572
Title: Evaluation of the Impact of a Personal and Domestic Hygiene Intervention on Lead Exposure in a Community Close to a Mine Dump
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Johannesburg (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Charlotte Mokoatle, Principal Investigator, University of Johannesburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Mining Intervention Study
Record Dates: First submitted 2022-02-18; First posted 2022-03-03 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Lead Poisoning; Lead Poison Children
Keywords: Lead; Lead exposure; Mine Dumps
MeSH Terms: conditions — Lead Poisoning

STUDY DESIGN:
Intervention Model Description: Participants are divided into two groups and one group is assigned to one household hygiene and an educational intervention which they apply and the impact of the intervention on lead exposure is assessed and the other group has no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The group that will receive the intervention to apply
  Interventions: Behavioral: Domestic Hygiene and household hygiene Intervention
- Control group (No Intervention): The group that will not receive the intervention

INTERVENTIONS:
Behavioral: Domestic Hygiene and household hygiene Intervention — A demonstration on the domestic hygiene intervention will be conducted where participants will be guided on optimal cleaning of windowsills, floors and other surfaces with water and detergent, and advised on appropriate method of cleaning. Participants will be provided with a package of cleaning materials (mop, bucket, detergent, hand wash liquid soap and cloth for wet dusting) which will be used during the demonstration, and retained by participants to facilitate sustainability of the intervention during and after the study. Participants will be further engaged in an educational discussion, with the aid of a specially designed educational pamphlet containing information about health effects potentially associated with dust lead exposure from mine dumps and the personal hygiene and domestic hygiene steps that may be followed to reduce dust lead exposure.
  Arms: Intervention group

SUMMARY:
The study evaluates the impact of a personal and domestic hygiene intervention on exposure to lead in a community close to a mine dump. A before and after intervention study will be conducted in a selected area to determine lead exposure levels and the reduction or not after application of the intervention.

DETAILED DESCRIPTION:
A before and after intervention study will be conducted with a control and intervention group, where data will be collected at the household (through questionnaire based interviews, floor and/or windowsill samples and soil samples collection) and individual level (through hand dust wipe sample collection). In phase one, both the control and intervention group will be interviewed, household floor and/or windowsill dust wipes will be taken, yard soil sample collected and hand dust wipe samples will be taken from children in participating households. After baseline data collection, participants will be allocated into either intervention or control group. The intervention group will participate in the domestic hygiene demonstration and educational discussion.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of one and five years

Exclusion Criteria:

* Children above 5 years

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 576 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Lead exposure level | Three months
  To detect a mean difference in change from baseline to follow-up of -0.5 μg/dL between the control and experimental group, with common standard deviation of 2 μg/dL

SECONDARY OUTCOMES:
Reference Lead exposure level | Three months
  A reference level of 5.0 μg/dL for public health intervention of exposure to lead

CONTACTS AND LOCATIONS:
Overall Officials: Makhutsisa C Mokoatle, Masters, Principal Investigator — University of Johannesburg; Vusumuzi Nkosi, PhD, Study Director — Medical Research Council, South Africa
Locations (1):
- Snake Park, Soweto, Johannesburg, Gauteng, South Africa

IPD SHARING:
Plan to Share IPD: Yes
All collected IDP to be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Through out the duration of the study up to a period of five years
Access Criteria: Only the research team will access IPD for capturing and analysis of covariance and descriptive statistics.

REFERENCES:
- [Derived] Mokoatle C, Mathee A, Street R, Nkosi V. A study protocol to evaluate the impact of a personal and domestic hygiene intervention on lead exposure in a community next to a mine dump. BMC Public Health. 2022 Jun 4;22(1):1123. doi: 10.1186/s12889-022-13439-8. PMID 35658916